CLINICAL TRIAL: NCT01778192
Title: A Randomized Prospective Trial Comparing Different Regimens of Polyethylene Glycol-based Lavage and Sodium Picosulphate With Magnesium Citrate in the Preparation of Patients for Colonoscopy
Brief Title: A Randomized Prospective Trial Comparing Polyethylene Glycol and Sodium Picosulphate With Magnesium Citrate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Woo-Jin Lee, fellow, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Korea University
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer; Colon Adenoma
Keywords: Bowel preparation; Polyethylene glycol; Sodium picosulphate
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Polyethylene Glycols; picosulfate sodium; magnesium citrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Same day PEG (Active Comparator): group 1 (same day PEG, N=50) received 4 L of PEG at 6 hours before procedure on the day of the colonoscopy
  Interventions: Drug: Polyethylene glycol
- split PEG (Active Comparator): group 2 (split PEG, N=50) received 2 L of PEG at 6:00 p.m the evening before colonoscopy and 2 L of PEG at 4-6 hours before procedure
  Interventions: Drug: Polyethylene glycol
- SPMC 2 (Active Comparator): group 3 (SPMC 2, N=50) received one sachet of SPMC at 6 p.m the evening before colonoscopy and another sachet of SPMC at 4-6 hours before procedure
  Interventions: Drug: Sodium picosulphate with magnesium citrate
- SPMC 3 (Active Comparator): group 4 (SPMC 3, N=50) received one sachet of SPMC at 6 p.m and the other sachet at 9 p.m the evening before colonoscopy and another sachet at 4-6 hours before procedure.
  Interventions: Drug: Sodium picosulphate with magnesium citrate

INTERVENTIONS:
Drug: Polyethylene glycol — -group 1 (same day PEG) received 4 L of PEG at 6 hours before procedure on the day of the colonoscopy
  Other Names: Colyte(Taejoon Pharmaceuticals, Seoul, Korea)
  Arms: Same day PEG
Drug: Polyethylene glycol — -group 2 (split PEG, N=50) received 2 L of PEG at 6:00 p.m the evening before colonoscopy and 2 L of PEG at 4-6 hours before procedure
  Other Names: Colyte(Taejoon Pharmaceuticals, Seoul, Korea)
  Arms: split PEG
Drug: Sodium picosulphate with magnesium citrate — -group 3 (SPMC 2) received one sachet of SPMC at 6 p.m the evening before colonoscopy and another sachet of SPMC at 4-6 hours before procedure
  Other Names: Picolight(Pharmbio korea, Seoul, Korea)
  Arms: SPMC 2
Drug: Sodium picosulphate with magnesium citrate — -group 4 (SPMC 3) received one sachet of SPMC at 6 p.m and the other sachet at 9 p.m the evening before colonoscopy and another sachet at 4-6 hours before procedure.
  Other Names: Picolight(Pharmbio korea, Seoul, Korea)
  Arms: SPMC 3

SUMMARY:
Adequate bowel cleansing is important for a completeness of colonoscopy and detection of colon polyps. Inadequate bowel preparation leads to longer duration of colonoscopy and obscured mucosal visualization resulting in missed lesions.

Bowel cleansing agents are simply classified into the large volume, iso-osmotic polyethylene glycol (PEG) based solutions or the small volume osmotically active agents, such as sodium picosulphate with magnesium citrate (SPMC).

There are rare reports that compare directly conventional polyethylene glycol (PEG) solution and sodium picosulphate with magnesium citrate (SPMC) for bowel preparation in korea.

The aim of this study is to compare the efficacy, safety, and tolerability of different regimens of SPMC and PEG solution.

DETAILED DESCRIPTION:
1. Study design: endoscopist-blinded, prospective, randomized controlled trial
2. Subjects

   1. Entry criteria: Male or female patients, aged between18 and 75 years undergoing elective outpatient colonoscopy were eligible for the study.
   2. Exclusion criteria:

   gastrointestinal obstruction or perforation, toxic megacolon, severe uncontrolled inflammatory bowel disease, previous colorectal resection, congestive heart failure, recent acute myocardial infarction or unstable angina, uncontrolled arterial hypertension, renal insufficiency with glomerular filtration rate < 60 ml/minute/1.73 m2, liver cirrhosis or ascites, pregnancy, lactation, and history of hypersensitivity to any bowel cleansing agents.
3. Sampling design: Consecutive recruitment of consenting patients
4. Variables Predictor

   1. group 1 (same day PEG) received 4 L of PEG at 6 hours before procedure on the day of the colonoscopy
   2. group 2 (split PEG) received 2 L of PEG at 6:00 p.m the evening before colonoscopy and 2 L of PEG at 4-6 hours before procedure
   3. group 3 (SPMC 2) received one sachet of SPMC at 6 p.m the evening before colonoscopy and another sachet of SPMC at 4-6 hours before procedure;
   4. group 4 (SPMC 3) received one sachet of SPMC at 6 p.m and the other sachet at 9 p.m the evening before colonoscopy and another sachet at 4-6 hours before procedure.
5. Primary Outcome: Quality of bowel preparation (Ottawa scale)
6. Secondary Outcome: Tolerability, palatability, side effect of the cleansing agents

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged between18 and 75 years undergoing elective outpatient colonoscopy were eligible for the study

Exclusion Criteria:

* gastrointestinal obstruction or perforation, toxic megacolon, severe uncontrolled inflammatory bowel disease, previous colorectal resection, congestive heart failure, recent acute myocardial infarction or unstable angina, uncontrolled arterial hypertension, renal insufficiency with glomerular filtration rate < 60 ml/minute/1.73 m2, liver cirrhosis or ascites, pregnancy, lactation, and history of hypersensitivity to any bowel cleansing agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
the quality of the bowel preparation using the Ottawa bowel preparation scale (OBPS) | 20 minutes
  Immediately following the colonoscopy, the endoscopist who were unaware of the preparation regimen scored the quality of the bowel preparation using the Ottawa bowel preparation scale (OBPS).

SECONDARY OUTCOMES:
Completeness of the bowel preparation | 30 minutes before the colonoscopy
  Patient compliance was recorded by checking the completeness of the prescribed preparation methods including bowel cleansing agent solution and recommended clear liquid.
the patient's tolerability | 30 minutes before the colonoscopy
  Patients were asked with questionnaires about the symptoms associated with the preparation to assess the patients' tolerability before the colonoscopy. Patients were asked whether they experienced any of the following : abdominal fullness, cramping, nausea, vomiting, sleep disturbance, and overall discomfort, and these symptoms were scored on a 5-point scale where 1 = "none", 2 = "mild", 3 = "moderate", 4 = "severe", and 5 = "very severe".
the side effects of the sodium picosulphate and magnesium citrate | 1 hour before the colonoscopy
  Biochemical measures detected outrange of serum electrolytes (sodium, potassium, chloride, calcium, magnesium, and phosphate), blood urea nitrogen, creatinine and serum osmolality only for the sodium picosulphate and magnesium citrate.
  Biochemical measurement was done done for the patients in the polyethylene glycol groups due to the well established safety date of the polyethylene glycol solutions.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Tae Jeen, Study Director — Division of Gastroenterology, Department of Internal Medicine, Korea University College of Medicine, Seoul, Republic of Korea; Eun Sun Kim, Principal Investigator — Division of Gastroenterology, Department of Internal Medicine, Korea University College of Medicine, Seoul, Republic of Korea; Woo Jin Lee, Principal Investigator — Division of Gastroenterology, Department of Internal Medicine, Korea University College of Medicine, Seoul, Republic of Korea
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine, Korea University College of Medicine, Seoul, South Korea